CLINICAL TRIAL: NCT07260318
Title: Acute Effects of Cricket Fast Bowling on Bone Turnover and Signaling Markers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Professor, Loughborough University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11201
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Health Adults
Keywords: Cricket; Fast bowling; Bone turnover; Stress injuries
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Bowling + Control (Experimental): Participants first perform the bowling trial, followed by the control trial, with a minimum interval of one week between the two trials.
  Interventions: Behavioral: Exercise
- Arm Control + Bowling (Experimental): Participants first perform the control trial, followed by the bowling trial, with a minimum interval of one week between the two trials.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — During the bowling trial, participants perform 8 sets of 6 deliveries (bowl at match intensity throughout), followed by 2-hour rest. Each set is interspersed by a 3-minute randomized fielding simulation. During the control trial, participants rest throughout instead of bowling.

SUMMARY:
The goal of this study is to investigate the acute effects of cricket fast bowling on the bone turnover and signaling markers in healthy young males.

The main question aims to answer:

• Does a single bout acute fast bowling change serum C-terminal telopeptide of type I collagen (CTX-I) and other bone turnover and signaling markers levels?

Participants complete both the bowling and control trials, with a minimum washout period of one week between trials. During each trial, blood samples are collected at three time points: pre-, immediately post, and 2-hour post bowling/rest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Aged 18 - 30
* Cricket fast bowlers (a ball speed of ~100kmh) playing for a university team or above, such as British Universities and Colleges Sport (BUCS) or University Centre of Cricketing Excellence (UCCE)
* Injury free for the last 3 months

Exclusion Criteria:

* Diagnosed with any disease or use of any medication that affects bone turnover
* Fracture experienced within the previous year/season

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum C-terminal telopeptide of type I collagen (CTX-I) concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum CTX-I concentration is measured using electrochemiluminescence immunoassay (ECLIA) and reported in nanograms per milliliter (ng/mL).

SECONDARY OUTCOMES:
Serum N-terminal propeptide of type I collagen (PINP) concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum PINP concentration is measured using electrochemiluminescence immunoassay (ECLIA) and reported in nanograms per milliliter (ng/mL).
Serum parathyroid hormone (PTH) concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum PTH concentration is measured using electrochemiluminescence immunoassay (ECLIA) and reported in picograms per milliliter (pg/mL).
Serum sclerostin concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum sclerostin concentration is measured using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Serum dickkopf Wnt signaling pathway inhibitor 1 (DKK1) concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum DKK1 concentration is measured using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Serum osteoprotegerin (OPG) concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum OPG concentration is measured using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Serum irisin concentration | Blood samples are collected at baseline, immediately after the bowling or the corresponding rest period, and 2 hours after the second blood sample collection.
  Serum irisin concentration is measured using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Bowling speed | Bowling speed is measured during the bowling trial.
  Bowling speed is measured using a radar gun during the 8 overs of bowling and reported in miles per hour (MPH).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavell, Principal Investigator — Loughborough University
Locations (1):
- Loughborough Univeristy, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No